CLINICAL TRIAL: NCT07186725
Title: Home-Based Under-Mattress Monitoring Device to Estimate Mandibular Advancement in Oral Appliance Therapy for Obstructive Sleep Apnea
Brief Title: Home-based Under Mattress Monitor for OSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Isabel Moreno Hay (Other)
Collaborators: American Academy of Dental Sleep Medicine (Unknown)
Responsible Party: Sponsor-Investigator, Isabel Moreno Hay, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 97445
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Obstructive Sleep Apnea (OSAS); Obstructive Sleep Apnea (SAOS)
Keywords: Mandibular Advancement; Sleep Apnea; Oral Appliance; Home-based; Obstructive Sleep Apnea; Home-based device
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Occlusal Splints

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Panthera DSAD mandibular advancement device users (Experimental): Participants of the study that have been referred to the Orofacial Pain Clinic by their sleep physician for the management of their obstructive sleep apnea with a mandibular advancement device.
  Interventions: Device: Under-mattress monitor; Device: level 3 Home Sleep Apnea Test; Device: Mandibular Advancement Device (MAD)

INTERVENTIONS:
Device: Under-mattress monitor — the under-mattress monitor will be used in conjunction with the Alice NightOne at the beginning and end of the study, in addition, the under-mattress monitor will be used daily during sleep with the intraoral device in situ
  Other Names: Sleeptracker-AI
Device: level 3 Home Sleep Apnea Test — Home sleep apnea test with Alice NightOne will be used for one day during sleep at the beginning and end of the study in conjunction with the Sleeptracker AI and the intraoral device.
  Other Names: Alice NightOne
Device: Mandibular Advancement Device (MAD) — CAD-CAM, US Food and Drug Administration (FDA)-approved MAD, duo-bloc, customized, titratable sleep appliance. Participants will return every 2 weeks to the Orofacial Pain (OFP) clinic to progressively titrate the MAD advancement as needed until the under-mattress monitor scores an AHI < 5
  Other Names: D-SADTM Panthera Dental

SUMMARY:
The aim of the study is to evaluate the effectiveness of the under-mattress monitoring device to aid in the titration process of a mandibular advancement device (MAD) for the management of obstructive sleep apnea (OSA). A secondary aim is to evaluate changes in subjective OSA symptoms and patient's satisfaction with MAD. A third aim is to analyze if there are differences between the sleep parameters recorded by the under-mattress monitor between responders and non-responders to MAD therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Obstructive Sleep Apnea demonstrated with a sleep study polysomnography or home sleep study (PSG or HSAT), manually scored by a sleep physician according to the 2017 American Academy of Sleep medicine scoring guidelines.
* Willingness to commute to the OFP clinic every 2 weeks during MAD titration period.
* Consent to partake in the study.

Exclusion Criteria:

* Diagnosis of central or mixed sleep apnea.
* Neurocognitive disease.
* Concomitant therapy with PAP therapy.
* Allergic to the appliance material (Polyamide 12).
* Presence of active dental decay, ill-fitting dental restorations, or crown to root ratio unfavorable.
* Inadequate English language comprehension.
* Lack of coordination or dexterity to insert/remove the MAD intraorally.
* Inability to tolerate digital dental impressions.
* Patients with concomitant diagnosed sleep disorders, including narcolepsy, restless leg syndrome, rapid eye movement sleep behavior disorder).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01-07 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in apnea-hypopnea index (AHI). | Baseline and post-intervention (approximately 12 weeks)
  Number of apneas and hypopneas per hour of sleep which is an indicator of severity of sleep apnea, (5< normal, 5-15 Mild, 15-30 moderate, <30 severe)
Change in minimum oxygen desaturation level | Baseline and post-intervention (approximately 12 weeks)
  The minimum O2 level percentage during treatment

SECONDARY OUTCOMES:
Change in Epworth Sleepiness Scale | Baseline and post-intervention (approximately 12 weeks)
  This scale measures daytime sleepiness. Scores range from 0-24. Higher scores indicate more severe daytime sleepiness.
Change in Quality of Life Scale | Baseline and post-intervention (approximately 12 weeks)
  Quality of life (15D questionnaire) with 15 question items with 5 alternatives in each. The scores range between 15 to 75 with 15 the best and 75 the worst quality of life.
Change in Fatigue Assessment Scale | Baseline and post-intervention (approximately 12 weeks)
  The scale consists of 10 questions about the characteristics of fatigue in the current daily routine. The scale scores range from 10-50, with higher score indicating higher level of fatigue.
Change in Pittsburgh Sleep Quality Index (PSQI) | Baseline and post-intervention (approximately 12 weeks)
  The PSQI is a 19-item questionnaire that includes seven areas of sleep quality and patterns in adults over the last month including the following components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, SDs, use of sleeping medications, and daytime dysfunction. Each item in the scale is scored from 0 to 3 scale (0 = no difficulty; 3 = severe difficulty). The scores are added to yield a global score ranging from 0 to 21 (0 = no difficulty; 21 = severe difficulties in all areas). A high total scale score indicates poor sleep quality.
Change in Snore Outcomes Survey (SOS) | Baseline and post-intervention (approximately 12 weeks)
  SOS consists of eight items related to the frequency, duration, severity, and consequences associated with sleep-disordered breathing and specifically snoring. Respondents use several Likert-type scales to answer questions regarding their snoring, with lower scores indicating more acute problems with SDB. Scores are normalized on a scale from 0 to 100.
Short Assessment of Patient Satisfaction | Post Intervention, approximately week 12
  Patient satisfaction with MAD will be measured by a 7-item questionnaire scored on a Likert type scale. Scores range from 7 to 35. Higher scores equate to greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Moreno Hay, DDS, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No